CLINICAL TRIAL: NCT05840536
Title: Efficacy and Tolerability of Combination Intravenous Diuretic Therapy Versus Intravenous Loop Diuretic Therapy Alone for the Treatment of Acute Decompensated Heart Failure
Brief Title: Combination Diuretic Therapy for Acute Decompensated Heart Failure
Acronym: COMBIND-HF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OchsnerHS
Record Dates: First submitted 2014-04-22; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Acute Decompensated Heart Failure
Keywords: heart failure; acute; diuretic; management; renal function; chlorothiazide; furosemide
MeSH Terms: conditions — Heart Failure | interventions — Furosemide; Chlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Diuretic Therapy (Experimental): Patients will receive lasix infusion starting at 5mg/hr along with a bolus dose of chlorothiazide 250mg at the initiation of the protocol. The lasix infusion can be titrated to 10mg after 12hrs based on volume of diuresis. This arm will also receive 250mg bolus doses of chlorothiazide every 12hrs for the duration of the study.
  Interventions: Drug: Furosemide plus Chlorothiazide; Drug: Furosemide
- Monotherapy Diuretic (Active Comparator): Patients will receive furosemide infusion at 5mg/hr along with an initial bolus dose of furosemide equal to twice their home oral dose. The furosemide infusion can be increased to 10mg/hr after 12hrs based on urine output. This arm will receive bolus doses of furosemide every 12hrs equal to twice their home oral dose until completion of the protocol.
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide plus Chlorothiazide — Patients will receive lasix infusion starting at 5mg/hr along with a bolus dose of chlorothiazide 250mg at the initiation of the protocol. The lasix infusion can be titrated to 10mg after 12hrs based on volume of diuresis. This arm will also receive 250mg bolus doses of chlorothiazide every 12hrs for the duration of the study.
  Intravenous (IV) lasix infusion at 5mg/hr plus IV boluses of diuril every 12 hrs.
  Other Names: Lasix plus Diuril
  Arms: Combination Diuretic Therapy
Drug: Furosemide — Patients will receive furosemide infusion at 5mg/hr along with an initial bolus dose of furosemide equal to twice their home oral dose. The furosemide infusion can be increased to 10mg/hr after 12hrs based on urine output. This arm will receive bolus doses of furosemide every 12hrs equal to twice their home oral dose until completion of the protocol.
  Other Names: Lasix

SUMMARY:
Patients with heart failure are often admitted to the hospital because they have accumulated excessive amounts of fluid, they become short of breath and congested with fluid. Removing the excess fluid is necessary to improve the patients symptoms and reduce the risk of being re-admitted to the hospital. Diuretics ("water pills") are often given through an IV to accelerate the fluid removal. Furosemide is commonly used for fluid removal, however some patients do not respond well to the medication. There are other diuretics available that can work in conjunction with furosemide and increase the rate of fluid removal. The other "water pills" have slightly different mechanisms of action in the body compared to furosemide and when combined they may increase fluid removal.

The investigators hypothesize that adding chlorothiazide to furosemide will result in quicker and more effective fluid removal in heart failure patients.

DETAILED DESCRIPTION:
The investigators will randomly assign patients to receive either furosemide alone or furosemide in combination with chlorothiazide when they are admitted to the hospital with acute heart failure and excessive volume.

All patients will be monitored for rate of fluid removal, improvement in symptoms, and side-effects of the medications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Decompensated Heart Failure - by at least 1 symptom (dyspnea, exercise intolerance, weight gain, edema) and at least 1 sign (chest x-ray (CXR), elevated brain natriuretic peptide (BNP), rales, elevated jugular venous pressure (JVP)).
* History of Congestion Heart Failure (CHF) with chronic loop diuretic use for at least the past 4 weeks
* Echocardiogram in the past 12 months (to document Ejection fraction (EF))

Exclusion Criteria:

* Chronic Kidney Disease (CKD) or Acute Kidney Injury (AKI) - Cr >2.5 mg/dL
* Ventricular assist device
* Cardiogenic shock
* Need for mechanical or vasopressor support on admission
* Significant co-morbidities: Chronic Obstructive Pulmonary Disease, pneumonia, pulmonary embolism
* History of pulmonary hypertension (PAH) (World Health Organization (WHO) group I primary PAH)
* Acute Ischemia / post-intervention (Coronary Artery Bypass Graft, Percutaneous Coronary Interventions) in the past 90 days

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Volume of Diuresis | During Index Hospitalization at 72 hours
  Total volume of urine output will be collected during the first 72 hours of admission.
Change in Serum Creatinine from Baseline | During Index Admission up to 120 hours
  Change in serum creatinine from baseline after 72 hours of diuresis

SECONDARY OUTCOMES:
Hypokalemia | From date of index hospitalization until 72 hours after diuresis
Electrolyte Disturbances | From date of index hospitalization until 72 hours after diuresis
  Magnesium, Phosphorous
Total Weight Loss | From date of index hospitalization until 72 hours after diuresis
Relief of Symptoms | From date of index hospitalization until 72 hours after diuresis
  Using the five-point Likert scale for dyspnea which ranges from 1-5 where the lower the score the better the outcome
Length of Stay | From date of index hospitalization until date of discharge from hospital, assessed up to 1 week
Potassium Replacement Requirements | From date of index hospitalization until date of discharge from hospital, assessed up to 1 week
Adverse Events | From date of index hospitalization until date of discharge from hospital, assessed up to 1 week
  Hypotension, dizziness, syncope, acute renal failure, arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T Campbell, MD, Study Director — Ochsner Heart and Vascular Institute; Stacy Mandras, MD, Principal Investigator — Ochsner Heart and Vascular Institute
Locations (1):
- Ochsner Heart and Vascular Institute, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Felker GM, Lee KL, Bull DA, Redfield MM, Stevenson LW, Goldsmith SR, LeWinter MM, Deswal A, Rouleau JL, Ofili EO, Anstrom KJ, Hernandez AF, McNulty SE, Velazquez EJ, Kfoury AG, Chen HH, Givertz MM, Semigran MJ, Bart BA, Mascette AM, Braunwald E, O'Connor CM; NHLBI Heart Failure Clinical Research Network. Diuretic strategies in patients with acute decompensated heart failure. N Engl J Med. 2011 Mar 3;364(9):797-805. doi: 10.1056/NEJMoa1005419. PMID 21366472
- [Background] Channer KS, McLean KA, Lawson-Matthew P, Richardson M. Combination diuretic treatment in severe heart failure: a randomised controlled trial. Br Heart J. 1994 Feb;71(2):146-50. doi: 10.1136/hrt.71.2.146. PMID 8130022
- [Background] Peacock WF, Costanzo MR, De Marco T, Lopatin M, Wynne J, Mills RM, Emerman CL; ADHERE Scientific Advisory Committee and Investigators. Impact of intravenous loop diuretics on outcomes of patients hospitalized with acute decompensated heart failure: insights from the ADHERE registry. Cardiology. 2009;113(1):12-9. doi: 10.1159/000164149. Epub 2008 Oct 17. PMID 18931492